CLINICAL TRIAL: NCT01245309
Title: Endometrial Injury Prior to Controlled Ovarian Stimulation (COH) in Women Undergoing In-vitro Fertilization in Women With Previous IVF Failure.
Brief Title: Endometrial Scratching Prior to Controlled Ovarian Stimulation (COH) in Women Undergoing In-vitro Fertilization With Previous IVF Failure
Acronym: ESICOHF
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Gibreel, Dr, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AG1001
Record Dates: First submitted 2010-11-19; First posted 2010-11-22 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2014-01

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- scratching (Experimental): endometrial scratching prior ivf cycle
  Interventions: Procedure: scratching; Procedure: A PLACEBO PROCEDURE
- PLACEBO (Placebo Comparator): PLACEBO PROCEDURE
  Interventions: Procedure: A PLACEBO PROCEDURE

INTERVENTIONS:
Procedure: scratching — endometrial scratching before COH in IVF
  Arms: scratching
Procedure: A PLACEBO PROCEDURE — A PLACEBO PROCEDURE

SUMMARY:
Scratching the linning of the womb before IVF cycle could increase the chances of having a baby after an IVF cycle.

DETAILED DESCRIPTION:
All women with history of RIF (as defined by ESHRE) and who wish to undertake another assisted conception treatment cycle are invited to participate in the trial. Women will be randomised to two arms; one undergoing endometrial sampling and control. Women in the experimental arm will be subjected to endometrial scrapping with Pipelle biopsy catheter two times; on days 21 and 26 of the cycle prior to the IVF index cycle and after initiation of the GnRHa in the long agonist protocol. Women in the control group will undergo a placebo procedure using the uterine sound on the same days of the cycle like women in the intervention group.

ELIGIBILITY:
Inclusion Criteria:

WOMEN WITH PREVIOUS IVF FAILURE UNDERGOING IVF TREATMENT

-

Exclusion Criteria:

* WOMEN>40 YEARS OLD WOMEN UNDERGOING THEIR FIRST IVF TREATMENT CYCLE

Max Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 500 (Actual)
Dates: Start 2010-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
live birth rate per woman | 9 months

SECONDARY OUTCOMES:
ongoing pregnancy rate | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Egypt